CLINICAL TRIAL: NCT02946034
Title: Safety, Efficacy, and Changes in Traditional and Novel Biomarkers of Kidney Function in Patients With Hepatitis C and Advanced Chronic Kidney Disease Treated With Abbvie Viekira Pak or Mavyret Regimen
Brief Title: Viekira Pak or Mavyret Treatment for Patient With Chronic Kidney Disease and Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Raymond Chung, Director, Hepatology, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001822
Record Dates: First submitted 2016-10-21; First posted 2016-10-26 (Estimated); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Chronic Kidney Disease; Chronic Hepatitis C
Keywords: CKD; HCV
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hepatitis C, Chronic | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Intervention Model Description: This a single-arm study. Initially, Viekira Pak was available through Abbvie. However, once Mavyret became available, it supplanted Viekira Pak as the study medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Viekira Pak ± ribavirin or Mavyret (Experimental): 12 week therapy with Viekira Pak ± ribavirin
  8 or 12 week therapy with Mavyret
  Interventions: Drug: Viekira Pak ± ribavirin; Drug: Mavyret

INTERVENTIONS:
Drug: Viekira Pak ± ribavirin — 12 weeks treatment with AbbVie Viekira Pak ± ribavirin
  Other Names: AbbVie 3D regimen
Drug: Mavyret — 8 or 12 weeks treatment with AbbVie Mavyret

SUMMARY:
Open-label experimental trial of 12 weeks of Viekira Pak treatment ± ribavirin or Mavyret for adults with chronic kidney disease and hepatitis C.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effect of paritaprevir/ritonavir, ombitasvir, dasabuvir (referred to as Viekira Pak) ± ribavirin or Glecaprevir / Pibrentasvir (referred to as Mavyret) for adults with advanced CKD with an estimated glomerular filtration rate (eGFR) less than 45ml/min that are infected with hepatitis C virus (HCV) genotype 1 and to determine the effect of treatment on traditional and novel markers of kidney function and cardiovascular disease risk in patients with advanced CKD. During the course of this prospective, single arm treatment trial, we will measure currently accepted markers of kidney function and novel biomarkers of CKD progression to determine if they improve with eradication of HCV.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 year of age
2. HCV genotype 1 ≥ 1000 IU/mL
3. 6. Estimated glomerular filtration rate 15-45mL/min/1.73m2 as estimated by CKD-Epi equation

Exclusion Criteria:

1. Pregnant or lactating females
2. Uncontrolled depression or psychiatric disease
3. History or presence of any form of cancer within 3 years of enrollment
4. Experiencing life-threatening cryoglobulinemic vasculitis requiring initiation of rituximab, steroids or plasmapheresis.
5. Uncontrolled cardiovascular or pulmonary disease
6. Experiencing symptoms attributed to uremia
7. Anticipated need to begin renal replacement therapy in the next 6 months
8. History of kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Results data will be shared with the study sponsor and publication of data is anticipated.

RESULTS

PARTICIPANT FLOW:
Groups:
- Viekira Pak ± Ribavirin or Mavyret: 12 week therapy with Viekira Pak ± ribavirin (2 patients)
  8 or 12 week therapy with Mavyret (8 patients)
Period: Overall Study
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Two patients received AbbVie Viekira Pak ± ribavirin, and eight patients received Abbvie Mavyret (glecaprevir/pibrentasvir).
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Hepatitis C genotype [Count of Participants; unit: Participants]
  Genotype 1a | 4
  Genotype 1b | 2
  Genotype 2 | 1
  Genotype 3 | 2
  Genotype 4 | 1
Baseline estimated glomerular filtration rate (eGFR) [Count of Participants; unit: Participants]
  60-89 mL/min/1.73m2 | 1
  30-59 mL/min/1.73m2 | 4
  <30 mL/min/1.73m2 | 5
Hypertension [Count of Participants; unit: Participants] | 10
Diabetes [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Urine Tumor Necrosis Factor (TNF)-Alpha From Baseline to Post-treatment
Description: Measure of novel biomarkers of incident and progressive CKD and liver disease to determine if eradication of HCV infection changes the measures of chronic inflammation associated with progressive end-organ disease.
  To calculate the average change, the difference between baseline values and the average of 12-weeks post treatment and 40-weeks post treatment were found for each patient. These differences were then averaged, as shown below.
Time Frame: 52 Weeks
Population: 2 patients did not have urine TNF-alpha tested at these timepoints.
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
Number analyzed (Participants) | 8
ng/g | -0.05 (0.61)

2. Primary Outcome: Average Change in Urine Interleukin (IL)-6 From Baseline to Post-treatment
Description: as for outcome 1
Time Frame: 52 weeks
Population: 2 patients did not have urine IL-6 tested at these timepoints.
Measure: Mean (Standard Deviation); unit: ng/g
Groups:
- Viekira Pak ± Ribavirin or Mavyret: 12 week therapy with Viekira Pak ± ribavirin
  8 or 12 week therapy with Mavyret
  Viekira Pak ± ribavirin: 12 weeks treatment with AbbVie Viekira Pak ± ribavirin
  Mavyret: 8 or 12 weeks treatment with AbbVie Mavyret
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
Number analyzed (Participants) | 8
ng/g | 5.73 (12.18)

3. Primary Outcome: Average Change in Plasma Tumor Necrosis Factor (TNF)-Alpha From Baseline to Post-treatment
Description: as for outcome 1
Time Frame: 52 weeks
Population: 2 patients did not have plasma TNF-alpha tested at these timepoints.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
Number analyzed (Participants) | 8
pg/mL | 6.67 (42.87)

4. Primary Outcome: Average Change in Plasma Interferon Gamma-induced Protein 10 (IP-10) From Baseline to Post-treatment
Description: as for outcome 1
Time Frame: 52 Weeks 52 Weeks 52 weeks
Population: 2 patients did not have plasma IP-10 tested at these timepoints.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
Number analyzed (Participants) | 8
pg/mL | -394.57 (657.80)

5. Primary Outcome: Average Change in Plasma Interferon (IFN)-Gamma From Baseline to Post-treatment
Description: as for outcome 1
Time Frame: 52 weeks
Population: 2 patients did not have plasma IFN-gamma tested at these timepoints.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
Number analyzed (Participants) | 8
pg/mL | 2.01 (29.57)

6. Primary Outcome: Average Change in Plasma Interleukin (IL)-6 From Baseline to Post-treatment
Description: as for outcome 1
Time Frame: 52 weeks
Population: 2 patients did not have plasma IL-6 tested at these timepoints.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
Number analyzed (Participants) | 8
pg/mL | -3.94 (11)

7. Secondary Outcome: Number of Patients Who Suffered Adverse Events Related to Study Drug (Safety and Tolerability)
Description: Safety and tolerability of Viekira Pak treatment in CKD patients will be assessed by number of patients who suffered adverse events (serious or otherwise) deemed to be related to study drug.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
Number analyzed (Participants) | 10
Participants | 4

8. Secondary Outcome: Number of Patients Who Had Sustained Virologic Response at 12-weeks (SVR12) Post-treatment (Efficacy of Treatment)
Description: Efficacy will be determined by negative HCV RNA viral load measured during the 12 week treatment period as well as 12 weeks after the last dose.
Time Frame: 24 weeks
Population: 2 patients did not have hepatitis C checked after 12-weeks post-treatment; thus, we cannot definitively determine that they achieved SVR12.
Measure: Count of Participants; unit: Participants
Groups:
- Viekira Pak ± Ribavirin or Mavyret: 12 week therapy with Viekira Pak ± ribavirin (2 patients)
  8 or 12 week therapy with Mavryet (8 patients)
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: Each patient was followed for one year after initiation of treatment.
Description: Adverse events data collection was done at each study visit.
Groups:
- Viekira Pak ± Ribavirin or Mavyret: 12 week therapy with Viekira Pak ± ribavirin (2 patients)
  8 or 12 week therapy with Mavyret (8 patients
Arm/Group | Viekira Pak ± Ribavirin or Mavyret
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viekira Pak ± Ribavirin or Mavyret (N=10)
Stroke (Nervous system disorders) | 1 (1) — Occurred 30 weeks post-treatment, was deemed not related to study drug.
Seizure (Nervous system disorders) | 1 (1) — Occurred 19 weeks post-treatment, was deemed not related to study drug.
Fall / loss of consciousness (Nervous system disorders) | 1 (1) — Occurred 22 weeks post-treatment, was deemed not related to study drug.
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Occurred 29 weeks post-treatment, was deemed not related to study drug.
Cryoglobulinemic glomerulonephritis (Renal and urinary disorders) | 1 (1) — Occurred week 2 of treatment, was deemed not related to study drug.
Heart block (Cardiac disorders) | 1 (1) — Occurred week 5 of treatment, deemed possibly related to study drug (digoxin interaction with Mavyret).
Hypertensive emergency (Cardiac disorders) | 1 (1) — Occurred 39 weeks post-treatment, was deemed not related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viekira Pak ± Ribavirin or Mavyret (N=10)
muscle pain in leg (Musculoskeletal and connective tissue disorders) | 1 (1) — Reported at week 12 visit, deemed not related to study drug.
anemia (Blood and lymphatic system disorders) | 1 (1) — Observed at week 12 visit, deemed not related to study drug.
fatigue (Nervous system disorders) | 3 (3) — For one patient, reported at week 8 visit, deemed possibly related to study drug. For another, reported at week 4 visit, deemed possibly related to study drug. For another, reported at week 2 visit, deemed possibly related to study drug.
cryoglobulinemia (Blood and lymphatic system disorders) | 1 (1) — Observed at week 1 visit, deemed not related to study drug.
slow ventricular response (Cardiac disorders) | 1 (2) — Observed at week 8 visit and 12-weeks post treatment, deemed not related to study drug.
high potassium (Renal and urinary disorders) | 1 (1) — Observed at week 1 of treatment, deemed not related to study drug.

LIMITATIONS AND CAVEATS:
Our study has several limitations. Our pilot trial was limited by the small number of patients enrolled. Additionally, two subjects were lost to follow-up, decreasing the power of our analysis comparing pre- and post-treatment kidney function and biomarkers. Thus, the analysis presented is descriptive in nature. The analysis is limited by the absence of a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT02946034/Prot_SAP_000.pdf